CLINICAL TRIAL: NCT04253600
Title: Understanding the Predictive Factors and the Neurocognitive Basis of Developmental Language Disorder Original Public Title (French) : Projet ELENA, Etude Sur le développement du Langage Chez l'ENfAnt. Public Title (English) : Study on Infants' Language Development
Brief Title: Understanding the Predictive Factors and the Neurocognitive Basis of Developmental Language Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ELENA
Record Dates: First submitted 2020-01-21; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Developmental Language Disorders; Language Development
Keywords: Developmental Language Disorders; Predictive factors; Neural correlates; Neurocognitive basis; Language development; Natural-sleep MRI protocol
MeSH Terms: conditions — Language Development Disorders | interventions — Dihydrolipoamide Dehydrogenase; Environment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI Acquisition (Other): This does not refer to any group intervention. At-risk and control children will take part in a natural-sleep MRI protocol.
  Interventions: Behavioral: Risk profile screening questionnaire; Procedure: Investigation of the neural correlates of DLD using Magnetic Resonance Imagery (MRI); Behavioral: Online investigation of predictive factors associated with DLD and LANCOM app development; Behavioral: Individual behavioral and cognitive assessment; Behavioral: Automated analysis of language development and environment

INTERVENTIONS:
Behavioral: Risk profile screening questionnaire — Families will be asked to complete a LimeSurvey questionnaire that aims at evaluating general risk profiles associated with DLD (e.g., no elevated risk, behavioral risk, environmental risk, familial risk), as well as our exclusion criteria (e.g., hearing deficit).
Procedure: Investigation of the neural correlates of DLD using Magnetic Resonance Imagery (MRI) — MRI data acquisition will take place during natural sleep in infants aged from 6 to 12 months. First, families will have to complete a security questionnaire to make sure that neither the children nor the accompanying parent have any known contraindication preventing the MRI session and that none of them is wearing any ferro-magnetic elements. Then, families will be welcomed in a calm and child-friendly environment where we will propose them some preparatory games known to facilitate sleep in children. MRI protocol will comprise structural and functional images and won't exceed 30 minutes.
Behavioral: Online investigation of predictive factors associated with DLD and LANCOM app development — Parents will be asked to complete a series of online questionnaires every six months. Questionnaires will be created on LimeSurvey and will include different questionnaires, scales, and observations that aim at evaluating children's development, and especially language development, as well as parental and environmental characteristics.
Behavioral: Individual behavioral and cognitive assessment — Individual cognitive and behavioral assessment will be scheduled once a year, around the child's birth date, and will comprise an extensive battery of standardized evaluation appropriate for the child's age. This individual evaluation will focus on several developmental aspects including language, psychomotor, behavioral and cognitive development, as well as executive and socio-emotional functioning, depending on the age of the children. Evaluations will be adapted to each child's specific profile, while respecting the following administration rules: (1) we will prioritize language development testing, (2) testing sessions will be adapted to each child's pace and possibilities, (3) if a child does not want to take part in the assessment, feels tired, or does not seem to be comfortable with the investigator, tests won't be administered.
Behavioral: Automated analysis of language development and environment — Following the individual assessment, families will be asked to record their child's language environment over a 2-days' timeframe using the LENA® device, a "small wearable device allowing for large-scale all-day audio recording and automated vocal analyses of speech segments". An automatic analysis of the recordings, performed by the LENA pro software algorithms, will provide amongst others, a direct and natural measure of the child's number of vocalizations, adult word counts, conversational turns, duration of exposure to electronic media versus to meaningful language. Data acquisition will take place once a year following our sample selection, with a required recording time per day ranging from 12 to 16 hours.

SUMMARY:
For most children, language acquisition might appear like an effortless phenomenon, mostly arising from informal daily interaction with their surrounding people. Despite an adequate learning environment however, some children encounter major difficulties in learning their native tongue and develop a Developmental Language Disorder (DLD). Although the existence of a multi-factorial etiology has seemed to reach an agreement, presumably combining genetic and environmental factors to some kind of neural disruption, the underlying mechanisms leading to DLD are, to date, poorly understood.

Many studies have attempted to identify risk factors and early predictors associated with the future development of a language impairment. However, despite the constant efforts to identify early markers able to differentiate between transient and persistent language difficulties, early detection of children who will be developing a DLD remains highly difficult, partially due to the lack of direct and ecological measures of early language and communication development. In addition research on the causal neural correlates of DLD is in its infancy, and often compromised by small sample sizes or analyses methods that lack anatomical specificity to determine the neural correlates of language impairment.

Hence, In order to improve early detection and, therefore, language intervention, this longitudinal research project aims at investigating the early predictive factors as well as the neurocognitive basis of DLD by means of an integrative, multi-dimensional, and multi-methodological approach. To substantially gain insight, this research ideally integrates risk factors at multiple different levels, including the cognitive, neurobiological, parental and environmental level. From a methodological perspective, we will combine direct and indirect behavioral methods with neuroimaging methods in order to propose an early predictive model of language development.

DETAILED DESCRIPTION:
The present research project can be divided into four main data collection steps. The first step concerns families' recruitment through a principle of population-based screening. Parents and/or caregivers of children aged from 0 to 18 months will be asked to complete a screening questionnaire that aims to evaluate families' general risk profile associated with the development of DLD. A subsample of at-risk and control families will be selected based on the screening phase for longitudinal follow-up. The second step consists of the investigation of the neural correlates of DLD by using a natural-sleep MRI protocol in infants of 6 to 12 months old. The third step concerns the evaluation of predictive factors leading to DLD using indirect measures based on digital assessment of language development, parental and environmental characteristics (i.e., parents will have to fill in online questionnaires every 6 months during a 3-year timeframe). This step will also be dedicated to the development of an application that aims at evaluating early development of language and communication (i.e., LANCOM app). Finally, the fourth step comprises additional in-depth investigation of DLD's predictive factors, by means of direct measures, including individual cognitive and behavioral assessment, as well as an automated analysis of the child's language environment using the Language ENvironment Analysis digital language processor recording device (LENA®). Data collection for this last step will take place once a year over the whole project's timeframe.

ELIGIBILITY:
Inclusion Criteria:

* Having a child, preferably aged from 0 to 12 months, and a maximum of 18 months at the time of recruitment
* Having French as (one of) mother tongue(s)

Exclusion Criteria:

* Severe sensory deprivation resulting in hearing and/or visual impairment (i.e., deafness, blindness) detected at birth
* Chromosomal abnormalities (e.g., Down syndrome, Turner syndrome, Williams syndrome)
* Phenylketonuria
* Cleft lips or palates

Max Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1500 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Environmental characteristics | From 6 months to 48 months of age
  Online questionnaires to be completed by parents and evaluating environmental characteristics of the child.
Parental characteristics | From 6 months to 48 months of age
  Online questionnaires to be completed by parents and evaluating parental characteristics of the child.
Children's behavioral characteristics (indirect measure) | From 6 months to 48 months of age
  Online questionnaires to be completed by parents, which aims at evaluating children's development, and in particular, their language development.
Cognitive and behavioral characteristics (direct measure) as assessed by standardized batteries of tests | From 1 year to 4 years of age
  Individual cognitive and behavioral assessment evaluating several developmental aspects including language, psychomotor, behavioral and cognitive development, as well as executive and socio-emotional functioning (e.g., EVALObb, EVALO2-6, WPPSI-IV). We will use batteries of neuropsychological standardized evaluation appropriate for the child's age.
Evaluation of children's language development and environment using the Language ENvironment Analysis digital language processor recording device (LENA) | From 1 year to 4 years of age
  Automated analysis of language development and environment using the LENA device. An automatic analysis of the recordings, performed by the LENA pro software algorithms, will provide amongst others, a direct and natural measure of the child's number of vocalizations, adult word counts, conversational turns, duration of exposure to electronic media versus to meaningful language.
Magnetic Resonance Imagery analyses | 6-12 months old
  Evaluation of neural correlates of DLD using structural (and functional) images. Children aged from 6 months to 12(-18) months will be scanned only once.

SECONDARY OUTCOMES:
Risk profiles analysis based on risk screening online questionnaire | 0-18 months old (at screening)
  Evaluation of different risk profiles associated with the development of DLD (e.g., family risk, environmental risk) based on a risk screening online questionnaire to be completed by the parents.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Institut de recherche en sciences psychologiques (IPSY, UCLouvain), Louvain-la-Neuve
  - Institute of NeuroScience (IoNS, UCLouvain), Woluwe-Saint-Lambert

IPD SHARING:
Plan to Share IPD: Yes
As part of the evaluation of neural correlates, participants have to indicate in the inform consent form, whether they allow the research team to share their data with other researchers or not. Only anonymized MRI data are susceptible to be shared with other researchers if families explicitly mentioned it on inform consent.
Time Frame: Not specified at this time
Access Criteria: Only for people affiliated to the research institute or after signing a data use agreement.